CLINICAL TRIAL: NCT05695625
Title: The Effect of Bilateral Erector Spina Plane Block on Postoperative Analgesia in Cesarean Section Under Spinal Anaesthesia
Brief Title: The Effect of Bilateral Erector Spina Plane Block on Postoperative Analgesia in Cesarean Section Under SpinalAnaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Ahmet Onat Bermede (Unknown); Süheyla Karadağ Erkoç (Unknown); Volkan Baytaş (Unknown); Bulut Varlı (Unknown); Hanife Asuman Uysalel (Unknown)
Responsible Party: Principal Investigator, Bengi Safak, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraU-CS-ESPB
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative
Keywords: Erector spina plane block; postoperative pain; obstetric analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB (Active Comparator): Spinal anesthesia + bilateral ESPB (total of 40 ml, %0.5 bupivacaine)
  Interventions: Other: Spinal anesthesia + bilateral erector spine plane block
- Group SA (Active Comparator): Only spinal anesthesia
  Interventions: Other: Spinal anesthesia

INTERVENTIONS:
Other: Spinal anesthesia + bilateral erector spine plane block — Intraoperative period: Spinal anesthesia was administered with 0.5% bupivacaine and fentanyl 12.5mcg at the level of L4-5 interspace in the sitting position. At the end of the surgery, patients were given a sitting position with the help of 2 people for USG-guided ESPB. The high-frequency linear USG probe was placed in the midline at T12 level, after the spinous process visualized, the transverse process was visualized by moving probe 3-4cm laterally. After confirming the location of the needle tip with 1-2ml hydrodissection, 10 ml bupivacaine + 10 ml salin was applied both right and left sides.
  Postoperative period: If patients' VAS value >4, 75mg diclofenac intramuscular was administered. After 30 mins if patients' VAS values >4, 1000mg paracetamol intravenously was administered.
  Arms: Group ESPB
Other: Spinal anesthesia — Intraoperative period: Spinal anesthesia was administered with 0.5% bupivacaine and fentanyl 12.5mcg at the level of L4-5 interspace in the sitting position.
  Postoperative period: If patients' VAS value >4, 75mg diclofenac intramuscular was administered. After 30 mins if patients' VAS values >4, 1000mg paracetamol intravenously was administered.
  Arms: Group SA

SUMMARY:
Acute pain after cesarean section (SC) can be variable. Untreated pain can affect patients' life quality. Currently regional nerve blocks are frequently used as a part of multimodal analgesia. Erector spina plane block (ESPB), a recently defined interfacial plane block, provides multisegmental analgesia by spreading to both ventral and dorsal branches of the spinal nerve roots in the cranio-caudal plane with a single injection. The aim of this study is to evaluate the effects of ESPB on postoperative pain, analgesic use and patient satisfaction in patients delivered by CS under spinal anesthesia.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most common surgical procedures in the world. Acute pain intensity after cesarean section can be variable, making difficult to predict pain severity. Untreated pain can affect patients' life quality. Currently regional nerve blocks are frequently used as a part of multimodal analgesia. Erector spina plane block (ESPB) is a recently defined interfascial plane block. As a result of ultrasound (USG) guided local anesthetic drug injection into the fascial plane between erector spina muscle and vertebral transverse process, multisegmental analgesia provided by spreading to the both ventral and dorsal branches of the spinal nerve roots in cranio-caudal plane with a single injection. The primary aim of this study was to evaluate the effects of bilateral ESPB on postoperative pain, using the visual analog scale (VAS) in patients delivered by CS under spinal anesthesia. The secondary aims of the study are to evaluate the effects of ESPB on analgesic drug use and patient satisfaction in the postoperative period.

116 pregnants, aged between 18-45 years, delivered by CS from May 2020 to June 2021 included the prospective, randomised, single centre study. Exclusion criteria were age under 18 years, over 45 years, body mass index (BMI) over 35 kg/m2, ASA status over III, multiple pregnancy, preeclampsia, bleeding diathesis, opioid use and allergy to drugs to be used in the study. Spinal anesthesia was administered with 0.5% bupivacaine and fentanyl 12.5mcg at the level of L4-5 interspace with 26G quincke spinal needle in the sitting position. At the end of the surgery, in ESPB group, patients were given a sitting position with the help of 2 people for USG-guided ESPB. The high-frequency linear USG probe was placed in the midline at T12 level, after the spinous process visualized, the transverse process was visualized by moving probe 3-4cm laterally. After confirming the location of the needle tip with 1-2ml hydrodissection, 10 ml bupivacaine + 10 ml salin was applied both right and left sides. At the postoperative 2, 4, 6, 12 and 24th hours, patients' rest, cough, movement, low back and headache VAS values, analgesic drug use, first analgesic use time and satisfaction were evaluated. ESPB spread level was evaluated with pin-prick at the 4-6th hours. The SPSS 11.5 program was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* between 18-45 years, pregnants delivered by CS from May 2020 to June 2021

Exclusion Criteria:

* age under 18 years, over 45 years, body mass index (BMI) over 35 kg/m2, ASA status over III, multiple pregnancy, preeclampsia, bleeding diathesis, opioid use and allergy to drugs to be used in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  VAS scores at 2, 4, 6, 12 and 24th hours. (VAS is an 11 point numeric scale ranges from 0 to 10. )

SECONDARY OUTCOMES:
Postoperative analgesic drug consumption | 24 hours
  Diclofenac consumption in the first 24 hours was measured.
Need for rescue analgesic | 24 hours
  The number of patients who required rescue analgesic in the first 24 hours and paracetamol consumption were recorded.
Number of patients with postoperative nausea-vomiting and need of antiemetic usage | 24 hours
  Number of patients with postoperative nausea-vomiting and need of antiemetic usage were recorded.
Patients' satisfaction | 24 hours
  At the postoperative 2, 4, 6, 12 and 24th hours patients' satisfaction was assessed using a descriptive verbal scale (11 point scale from 0 to 10. 0: not satisfied, 10: very satisfied).
First analgesic using time, first mobilization time, hospitalization time | Postoperative 4 days on an average
  Postoperative first analgesic using time, first mobilization time and hospitalization time were recorded.
ESPB spread level | 4-6th hours
  The range of sensory block level in ESPB group was evaluated as dermatomal after the effect of spinal anesthesia passed, at 4-6th hours with pin-prick test.

CONTACTS AND LOCATIONS:
Overall Officials: Bengi Şafak, Principal Investigator — Ankara University
Locations (1):
- Bengi Şafak, Ankara, Turkey (Türkiye)